CLINICAL TRIAL: NCT01852942
Title: Reversing Tissue Fibrosis to Improve Immune Reconstitution in HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1111M06585; 13-3613 (Other: Hennepin County Medical Center); U01AI105872 (NIH)
Record Dates: First submitted 2012-02-20; First posted 2013-05-14 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: HIV Infection; HIV Infections
Keywords: Infection; HIV 1; HIV; Losartan; Fibrosis; Immune Activation; Immune Reconstitution
MeSH Terms: conditions — HIV Infections; Infections; Fibrosis | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan (Experimental)
  Interventions: Drug: Losartan
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Participants will start with 50 mg of losartan by mouth daily. The dose will be increased to 100 mg by mouth daily after 14 days. The maximal tolerable dosage (up to 100mg by mouth daily) will be continued for a total of 30 months.
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo — one tablet by mouth daily
  Arms: Sugar Pill

SUMMARY:
This study was designed to test the hypothesis that treatment of HIV infected subjects with losartan, an agent with specific anti-inflammatory and anti-fibrotic actions, will:

1. reverse existing lymphoid tissue fibrosis,
2. restore lymphoid tissue architecture,
3. increase the number and improve the function of peripheral and lymphatic CD4 T cells,
4. decrease levels of systemic immune activation (IA),
5. decrease size of the HIV reservoir, and
6. be safe and well tolerated.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial of 50 HIV-1 infected individuals on stable ART randomized in a 1:1 ratio to losartan (50 mg orally daily titrated to 100 mg daily) vs placebo for 30 months. We plan to enroll a total of 63 HIV infected subjects to ensure that 50 complete the protocol. All HIV infected subjects will undergo biopsies of inguinal lymph node (LN) and gut associated lymphatic tissue (GALT) for primary endpoint analysis at baseline, 12 and 30 months after study enrollment. Blood will be collected at least quarterly throughout the study and an intensive blood pharmacokinetic (PK) study will be conducted at month 1. All HIV infected subjects will be vaccinated with the quadrivalent human papillomavirus (HPV) vaccine at months 23, 25 and 29.5 to measure immune function. 5 HIV uninfected control subjects will also be enrolled.

The primary endpoint is to determine the impact of losartan on lymphoid tissue fibrosis in HIV infected, ART treated adults. This will be determined by measuring the amount of collagen deposition in lymphoid tissues and the integrity of the FRCn using immunohistochemistry (IHC) and quantitative image analysis (QIA).

ELIGIBILITY:
HIV infected participants:

1. Inclusion Criteria:

   Participants must meet all of the following inclusion criteria to participate in this study:
   * HIV-1 infected.

     -≥ 18 years of age.
   * Baseline peripheral CD4+ T cell count 200-600 cells/mm3 for at least two measures over the 6 months prior to study enrollment.

     -≥ 12 months of stable ART, defined as use of a given drug regimen without disruption lasting ≥ 1 week in the period leading up to study enrollment.
   * HIV viral load (VL) < 50 copies/mL for at least two consecutive measures over the 6 months prior to study enrollment.
   * No contraindication to proposed study procedures.
   * Women of child-bearing potential must be willing to use a form of effective contraception for the duration of the study. Effective contraception includes hormonal injection, implant or oral medication, IUD, diaphragm, or cervical cap with spermicide. Condoms cannot be used as the sole form of contraception.
2. Exclusion Criteria: Participants meeting any of the following exclusion criteria at baseline will be excluded from study participation:

   * Use of any immunomodulator within the 12 months prior to study enrollment. An immunomodulator for the purposes of this study is defined as a drug known to either diminish or augment a patient's immune system. Examples of these include, but are not limited to, systemic corticosteroids (use of topical steroids will be permitted), TNF-inhibitors, rituximab, cyclophosphamide, abatacept,cyclosporine, azathioprine, 6-mercaptopurine, methotrexate, sulfasalazine, cyclosporine, tacrolimus,sirolimus, and intravenous immune globulin.
   * Current use of an ARB or ACEi.
   * Current use of rifaximin, fluconazole or lithium given potential for drug interactions with losartan.
   * Prior reaction or intolerance to an ARB or ACEi.
   * Prior diagnosis of a chronic inflammatory disease with serologic or clinical evidence as diagnosed by a primary care physician or specialist. Examples of these include, but are not limited to, systemic lupus erythematosus, rheumatoid arthritis, scleroderma, Sjogren's syndrome, mixed connective tissue disease, psoriasis, polymyositis, dermatomyositis, vasculitis, sarcoidosis, Wegener's granulomatosis, giant cell arteritis, polyarteritis nodosa, gastrointestinal pemphigoid, eosinophilic colitis, Crohn's disease, ulcerative colitis, autoimmune hepatitis, and hepatitis C.
   * Prior diagnosis of a connective tissue disease with genetic, serologic or clinical evidence as diagnosed by a primary care physician or specialist (Marfan's syndrome, Ehlers-Danlos syndrome).
   * Baseline blood pressure < 110/70.
   * Estimated Glomerular Filtration Rate (eGFR) of < 30ml/min/1.73 m2 within 4 weeks of study initiation or history of advanced renal disease.
   * AST and/or ALT > 3 times the upper limit of normal within 4 weeks of study enrollment.
   * Potassium > 5.0 within 4 weeks of study enrollment.
   * Pregnancy.
   * In women of childbearing age, unwillingness to use birth control for the duration of the study.
   * Breast feeding.
   * Prior vaccination with an HPV vaccine, including Cervarix (GlaxoSmithKline) or Gardasil (Merck).
   * History of hypersensitivity or severe allergic reactions to yeast.

HIV-uninfected:

1. Inclusion Criteria

   Participants must meet all of the following inclusion criteria to participate in this study:
   * HIV uninfected.

     -≥ 18 years of age.
   * No contraindication to proposed study procedures.
2. Exclusion Criteria: Participants meeting any of the following exclusion criteria at baseline will be excluded from study participation:

   * Use of any immunomodulator within the 12 months prior to study enrollment (as defined above).
   * Current use of an ARB or ACEi.
   * Prior diagnosis of a chronic inflammatory disease with serologic or clinical evidence (as defined above).
   * Prior diagnosis of a connective tissue disease with genetic, serologic or clinical evidence as diagnosed by a primary care physician or specialist (Marfan's syndrome, Ehlers-Danlos syndrome).
   * Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Division of Infectious Diseases, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan: Losartan: We will start with 50 mg of losartan by mouth daily. We will increase the dosage to 100 mg by mouth daily after 14 days. The maximal tolerable dosage (up to 100mg by mouth daily) will be continued for a total of 30 months.
Period: Overall Study
Arm/Group | Losartan | Sugar Pill
Started | 25 | 27
Completed | 20 | 21
Not Completed | 5 | 6
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Sugar Pill | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11) | 50 (11) | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 25 | 26 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 11 | 12
  White | 19 | 14 | 33
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Collagen Deposition in LT
Description: The Impact of Losartan Treatment on Lymphoid Tissue (LT) Fibrosis will be determined by measuring the amount of collagen deposition in LT using immunohistochemistry (IHC) and quantitative image analysis (QIA). LT will be obtained at baseline, month 12 and month 30.
Time Frame: 30 months
Population: Some participant data was left out of this analysis due to sample quality.
Measure: Mean (Standard Deviation); unit: percent area
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 12 | 13
percent area
  12 months | 34.866 (9.3914) | 31.02 (5.6795)
  30 months | 30.8925 (9.4894) | 29.4492 (6.2988)

2. Primary Outcome: Integrity of the Fibroblastic Reticular Cell Network (FRCn)
Description: The Impact of Losartan Treatment on Lymphoid Tissue (LT) Fibrosis will be determined by measuring the Integrity of the fibroblastic reticular cell network (FRCn) using immunohistochemistry (IHC) and quantitative image analysis (QIA). LT will be obtained at baseline, month 12 and month 30.
Time Frame: 30 months
Population: This measure was planned at the time of registration, however it was not collected during the course of the trial. This data is not able to be reported.
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Frequency of CD4+ T Cells
Description: Impact of losartan on immune reconstitution and function will be determined by frequency of CD4+ T cells in LT using IHC.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Frequency TUNEL+CD3+CD8+ T Cells
Description: Impact of losartan on immune reconstitution and function will be determined by frequency of TUNEL+CD3+CD8+ T cells in LT using IHC.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Frequency of Cells Expressing TGF-beta and Lymphotoxin-beta
Description: Impact of losartan on immune reconstitution and function will be determined by frequency of cells expressing TGF-beta and lymphotoxin-beta in LT using IHC.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Serum Concentration of IL-7
Description: Impact of losartan on immune reconstitution and function will be determine by serum concentrations of IL-7 measured with ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Serum Concentration of TGF-beta
Description: Impact of losartan on immune reconstitution and function will be determine by serum concentrations of TGF-beta measured with ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Immune Response to HPV Vaccination
Description: Impact of losartan on immune reconstitution and function will be determine by measuring the immune response to HPV vaccination using flow cytometry to identify cells stimulated by specific HPV peptides.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Frequency of Activated T-cell Populations - Immunofluorescent Staining
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the frequency of activated T-cell populations (specifically CD3+CD4+CD38+, CD3+,CD8+CD38+,CD4+Ki67+ and CD8+Ki67+ T cells) in LT using immunofluorescence staining
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percent of Activated T Cells in PBMCs - Flow Cytometry
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the percentage of activated T cells in peripheral blood mononuclear cells (PBMCs) using flow cytometry.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percent of Activated Macrophages in PBMCs - Flow Cytometry
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the percentage of activated macrophages in peripheral blood mononuclear cells (PBMCs) using flow cytometry.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percent of Activated Dendritic Cells in PBMCs - Flow Cytometry
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the percentage of activated dendritic cells in peripheral blood mononuclear cells (PBMCs) using flow cytometry.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percent of Activated T Cells in LT - Flow Cytometry
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the percentage of activated T cells in lymphoid tissues (LT) using flow cytometry.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percent of Activated Macrophages in LT - Flow Cytometry
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the percentage of activated macrophages in lymphoid tissues (LT) using flow cytometry.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percent of Activated Dendritic Cells in LT - Flow Cytometry
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the percentage of activated dendritic cells in lymphoid tissues (LT) using flow cytometry.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Intracellular Concentration of IL-17 in PBMCs
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine IL-17 in PBMCs using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Intracellular Concentration of IFNg in PBMCs
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine IFNg in PBMCs using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Intracellular Concentration of IL-2 in PBMCs
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine IL-2 in PBMCs using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Intracellular Concentration of TNF in PBMCs
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine TNF in PBMCs using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Intracellular Concentration of IL-10 in PBMCs
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine IL-10 in PBMCs using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Intracellular Concentration of GM-CSF in PBMCs
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine GM-CSF in PBMCs using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Intracellular Concentration of IL-17 in LT
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine IL-17 in lymphoid tissue (LT) using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Intracellular Concentration of IFNg in LT
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine IFNg in lymphoid tissue (LT) using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Intracellular Concentration of IL-2 in LT
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine IL-2 in lymphoid tissue (LT) using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Intracellular Concentration of TNF in LT
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine TNF in lymphoid tissue (LT) using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Intracellular Concentration of IL-10 in LT
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine IL-10 in lymphoid tissue (LT) using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Intracellular Concentration of GM-CSF in LT
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the intracellular levels of the inflammatory cytokine GM-CSF in lymphoid tissue (LT) using cytokine staining.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Plasma Concentration of LPS
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of LPS by ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Plasma Concentration of sCD14
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of sCD14 by limulus assay.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Plasma Concentration of I-FABP
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of I-FABP using ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Plasma Concentration of IL-1b
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of IL-1b using ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Plasma Concentration of IL-1RA
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of IL-1RA using ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Plasma Concentration of IL-6
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of IL-6 using ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Plasma Concentration of TNF
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of TNF using ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Plasma Concentration of Amyloid A
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of amyloid A using ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Plasma Concentration of CRP
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of CRP using ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Plasma Concentration of D-dimer
Description: The Impact of Losartan on Immune Activation in HIV Infected, Treated Individuals will be determined by measuring the plasma concentration of D-dimer using ELISA.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Frequency of HIV RNA+ and DNA+ Cells in LN - Radiolabeled ISH
Description: The Potential for Losartan to Reduce the Size of the Viral Reservoir will be assessed by determining the frequency of HIV RNA+ and DNA+ cells in LN using radiolabeled in situ hybridization (ISH).
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Frequency of HIV RNA+ and DNA+ Cells in LN - RNAscopeTM in Situ Technology
Description: The Potential for Losartan to Reduce the Size of the Viral Reservoir will be assessed by determining the frequency of HIV RNA+ and DNA+ cells in LN using RNAscopeTM in situ technology.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Frequency of HIV RNA+ and DNA+ Cells in GALT - Radiolabeled in Situ Hybridization (ISH)
Description: The Potential for Losartan to Reduce the Size of the Viral Reservoir will be assessed by determining the frequency of HIV RNA+ and DNA+ cells in GALT radiolabeled in situ hybridization (ISH).
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Frequency of HIV RNA+ and DNA+ Cells in GALT - RNAscopeTM in Situ Technology
Description: The Potential for Losartan to Reduce the Size of the Viral Reservoir will be assessed by determining the frequency of HIV RNA+ and DNA+ cells in GALT using RNAscopeTM in situ technology.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Concentration of Losartan and Antiretrovirals (ARVs)
Description: Potential Drug-drug Interactions Between Losartan and Antiretrovirals (ARVs) will be assessed by measuring levels of ARVs and losartan in plasma and peripheral blood mononuclear cells (PBMCs).
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Intracellular Concentration of Losartan and Antiretrovirals (ARVs)
Description: Potential Drug-drug Interactions Between Losartan and Antiretrovirals (ARVs) will be assessed by measuring intracellular concentration of losartan and ARVs in lympoidtissue.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

44. Other Pre Specified Outcome: Frequency of Dendritic Cell and CD4 T Cell Interactions With the FRCn
Description: As an exploratory endpoint, we will determine the impact of losartan on frequency of dendritic cell and CD4 T cell interactions with the FRCn. This will be determined using two-photon microscopy in sections on LN obtained from study subjects. Given that this is an exploratory endpoint, these assays will be performed in a subset of subjects (5 losartan treated, 2 placebo treated and 5 HIV uninfected controls).
Time Frame: 30 months
Population: This exploratory endpoint was not analyzed and data are not available to be reported.
Arm/Group | Losartan | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Losartan | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 1/25 | 1/27
Serious Adverse Events (participants affected / at risk) | 2/25 | 6/27
Other Adverse Events (participants affected / at risk) | 25/25 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=25) | Sugar Pill (N=27)
Hospitalization for Chemotherapy (General disorders) | 1 (1) | 0 (0)
Hospitalization for Illness (General disorders) | 1 (1) | 5 (6)
Hospitalization for Surgery (General disorders) | 1 (1) | 5 (5)
Unintentional Weight Loss (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=25) | Sugar Pill (N=27)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (10)
Headache (General disorders) | 3 (3) | 2 (2)
Orthopedic injury (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Neuro-syphillis diagnosis (Infections and infestations) | 1 (1) | 0 (0)
Eye watering (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (9)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Arm pain/numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cold/flu symptoms (General disorders) | 2 (2) | 5 (5)
Toothache (General disorders) | 0 (0) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 2 (2) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (General disorders) | 1 (1) | 0 (0)
Light-headedness (General disorders) | 3 (3) | 1 (1)
Pustular node (General disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Jock itch (General disorders) | 1 (1) | 0 (0)
Sciatica, worsened (General disorders) | 2 (2) | 1 (1)
Neuropathy, worsened (Nervous system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 3 (3) | 1 (1)
Infected scatch (Infections and infestations) | 1 (1) | 0 (0)
Gas, belching (Gastrointestinal disorders) | 2 (3) | 1 (1)
Food poisoning (Infections and infestations) | 0 (0) | 1 (1)
Brain aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Pain/swelling at incision site (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Elevated blood glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Sinus infection (Infections and infestations) | 2 (2) | 2 (4)
Restless leg syndrome diagnoses (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mild sleep apnea (General disorders) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Liver cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fatigue/sluggishness (General disorders) | 6 (7) | 0 (0)
"Tight" feeling in nose and throat (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (5)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dry eyes (Eye disorders) | 1 (1) | 0 (0)
Dry mouth/cotton mouth (General disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign prostate hypertrophy (General disorders) | 0 (0) | 1 (1)
Night sweats (General disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Abdominal pain (General disorders) | 3 (3) | 0 (0)
Kidney stones (Renal and urinary disorders) | 1 (1) | 1 (1)
Fainting episode (General disorders) | 1 (1) | 0 (0)
Blood in stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
High blood pressure (General disorders) | 0 (0) | 3 (3)
Hot water burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bump at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Red, swollen area at drug injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sinus pain/congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Sores on gums (General disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Pinched nerve (Nervous system disorders) | 1 (1) | 0 (0)
Flu vaccine reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 2 (2)
Unknown weight loss (General disorders) | 1 (1) | 0 (0)
Borborygmus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloody nose (General disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 1 (1)
Numbness in hand (Nervous system disorders) | 0 (0) | 1 (1)
Heart burn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Groin pain (General disorders) | 0 (0) | 2 (2)
Heart palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Blastocis hominus (Infections and infestations) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Itchy rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Elevated creatinine (General disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Foot callus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Increased acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Bilateral foot pain (General disorders) | 0 (0) | 1 (1)
Microdiscectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Giardia (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (10) | 0 (0)
Colon polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 2 (2)
Temporal mandibular joint pain (General disorders) | 0 (0) | 1 (1)
Seasonal allergies (Immune system disorders) | 0 (0) | 1 (1)
Sleep disturbance (General disorders) | 0 (0) | 1 (1)
Rectal pain (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Increased viral load (Infections and infestations) | 0 (0) | 1 (1)
Excision of anal lesion (Surgical and medical procedures) | 0 (0) | 1 (1)
Multiple sclerosis flare-up (General disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cold sore (General disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (General disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toe infection (Infections and infestations) | 0 (0) | 1 (1)
Loss of consciousness during blood draw (General disorders) | 1 (2) | 0 (0)
Conjuctivitis (Eye disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Low blood pressure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sore throat (General disorders) | 2 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT01852942/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT01852942/ICF_001.pdf